CLINICAL TRIAL: NCT01375660
Title: Vitamin D Deficiency and Treatment in Male Veterans at Risk for Diabetes
Brief Title: D Vitamin Intervention in VA
Acronym: DIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CLIN-001-10S
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Results first posted 2015-02-05 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Impaired Fasting Glucose; Impaired Glucose Tolerance; Vitamin D Insufficiency
Keywords: Vitamin D; Glucose intolerance; African American men
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Placebo Comparator): Placebo: One capsule weekly
  Interventions: Drug: Placebo
- Arm 2 (Experimental): 50K vitamin D2: One capsule weekly
  Interventions: Drug: 50K vitamin D2

INTERVENTIONS:
Drug: Placebo — Supplement of vitamin D 400 units provided to all subjects, in addition Arm 1 will get placebo and Arm 2 will get D2 50K
  Arms: Arm 1
Drug: 50K vitamin D2 — Supplement of vitamin D 400 units provided to all subjects, in addition Arm 1 will get placebo and Arm 2 will get D2 50K
  Arms: Arm 2

SUMMARY:
This study will supplement African American male (AAM) veterans at risk for diabetes and newly diagnosed T2DM with vitamin D (low or higher dose) and evaluate whether vitamin D helps to improve early markers of diabetes. The study will be done at Veteran Administration Medical Center in Chicago.

DETAILED DESCRIPTION:
The goal of this randomized clinical trial (RCT) is to determine vitamin D efficacy and safety for improving early markers of T2DM in African American male (AAM) veterans at risk for T2DM (n=205, duration 12 months).

The primary outcome will be change in oral glucose insulin sensitivity (OGIS). The secondary outcomes will include various parameters of glucose metabolism and other biomarkers.

Analysis based on primary and secondary goal as well as predetermined levels of A1C, OGTT and 25OHD at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Veterans at Jesse Brown VA Medical Center (JBVAMC) only

* Male
* African American race
* Age 35-85 years
* BMI 28-39.9 kg/m2
* Stable weight (+/- 10%) for at least 3 months prior to study entry
* FPG 95 - 125 mg/dl
* A1C 5.7 - 6.4%
* Circulating 25OHD 5.0 - 29.9 ng/ml
* Subjects who take ergocalciferol are allowed in the study after a washout period 1 3 month.
* Subjects who take vitamin D supplements other than ergocalciferol are allowed in the study as long as total dose is no more than 600 IU/day (including MVI and calcium plus D supplements).
* Non-diabetic subjects who are diagnosed with T2DM during screening (A1C 6.5-7%) or after randomization are allowed to continue if they follow lifestyle intervention and do not need to take anti-diabetic medications.

Exclusion Criteria:

* Subjects with T2DM
* Weight gain or loss of more than 10% within 3 months prior to the study entry
* History of kidney stones, hyperparathyroidism, sarcoidosis or hypercalcemia
* A1C >7%.
* Very low 25OHD levels (<5 ng/ml) and/or the presence of a physical consequence of very low vitamin D levels (hypocalcemia, hypophosphatemia, proximal muscle weakness)
* Chronic kidney disease (CKD) stage 4 and 5
* Problems that in the judgment of PI may be associated with the risk to the subject or non-compliance
* Subjects who take vitamin D supplements and not willing to go through washout period for ergocalciferol or to take no more than 600 IU/day of total vitamin D supplements
* History, clinical manifestations or medications of significant metabolic, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, urological, neurological, psychiatric/ psychological disorders, or social circumstances which in the opinion of the investigator would be expected to interfere with the study or increase risk to the subject
* Non-diabetic subjects who are diagnosed with T2DM after randomization and need to take anti-diabetic medications are brought for the final visit

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena I. Barengolts, MD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

REFERENCES:
- [Derived] Ciubotaru I, Green SJ, Kukreja S, Barengolts E. Significant differences in fecal microbiota are associated with various stages of glucose tolerance in African American male veterans. Transl Res. 2015 Nov;166(5):401-11. doi: 10.1016/j.trsl.2015.06.015. Epub 2015 Jul 8. PMID 26209747
- [Derived] Eisenberg Y, Mohiuddin H, Cherukupally K, Zaidi H, Kukreja S, Barengolts E. Similarities and differences between patients included and excluded from a randomized clinical trial of vitamin D supplementation for improving glucose tolerance in prediabetes: interpreting broader applicability. Trials. 2015 Jul 15;16:306. doi: 10.1186/s13063-015-0812-0. PMID 26174313
- [Derived] Barengolts E, Manickam B, Eisenberg Y, Akbar A, Kukreja S, Ciubotaru I. EFFECT OF HIGH-DOSE VITAMIN D REPLETION ON GLYCEMIC CONTROL IN AFRICAN-AMERICAN MALES WITH PREDIABETES AND HYPOVITAMINOSIS D. Endocr Pract. 2015 Jun;21(6):604-12. doi: 10.4158/EP14548.OR. Epub 2015 Feb 25. PMID 25716637

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited among African American Male veterans coming for medical care to Jesse Brown VA Medical Center in Chicago between May 2011 and December 2012.
Groups:
- Placebo: supplement of vitamin D 400 units provided to all subjects in addition to placebo.
- 50K Vitamin D2: supplement of vitamin D 400 units provided to all subjects in addition to 50K vitamin D2.
Period: Overall Study
Arm/Group | Placebo | 50K Vitamin D2
Started | 102 | 103
Completed | 86 | 87
Not Completed | 16 | 16

BASELINE CHARACTERISTICS:
Groups:
- 50K Vitamin D2: Supplement of vitamin D 400 units provided to all subjects in addition to D2 50K.
- Total: Total of all reporting groups
Arm/Group | Placebo | 50K Vitamin D2 | Total
Number analyzed (Participants) | 86 | 87 | 173
Age, Customized [Number; unit: participants]
  35-85 Years | 86 | 87 | 173
Sex/Gender, Customized [Number; unit: participants]
  Male | 86 | 87 | 173
Race/Ethnicity, Customized [Number; unit: participants]
  African American Male Veterans | 86 | 87 | 173
Region of Enrollment [Number; unit: participants]
  United States | 86 | 87 | 173
BMI [Mean (Standard Deviation); unit: Kg/m2] | 31.5 (2.4) | 32.4 (2.9) | 31.9 (2.65)
HbA1c [Mean (Standard Deviation); unit: Percentage of A1C] | 6.1 (0.20) | 6.1 (0.26) | 6.1 (0.26)
Vit D [Mean (Standard Deviation); unit: ng/ml] | 14.0 (4.8) | 14.7 (4.7) | 14.3 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Oral Glucose Insulin Sensitivity (OGIS)
Description: Oral glucose insulin sensitivity = index of insulin sensitivity, higher index means higher insulin sensitivity. Low insulin sensitivity means high insulin resistance and high risk of type 2 diabetes mellitus. It is calculated by a special formula using insulin and glucose measured in Oral Glucose Tolerance test.
  The primary outcome was the change in oral glucose insulin sensitivity (OGIS, from oral glucose tolerance test) after 12 months of treatment calculated as OGIS at 12-months minus OGIS baseline.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ml/min/m^2 of body surface area
Arm/Group | Placebo | 50K Vitamin D2
Number analyzed (Participants) | 86 | 87
ml/min/m^2 of body surface area | -16.0 (55.83) | 7.8 (56.02)
Statistical Analysis 1: Comparison: Placebo vs 50K Vitamin D2; Test type: Superiority or Other; p = 0.026, ANOVA

2. Secondary Outcome: Change in HbA1c From Baseline at 12 Months
Time Frame: Baseline and 12 Months
Measure: Mean (Standard Deviation); unit: percentage of A1C
Arm/Group | Placebo | 50K Vitamin D2
Number analyzed (Participants) | 86 | 87
percentage of A1C | 0.01 (0.21) | -0.01 (0.18)
Statistical Analysis 1: Comparison: Placebo vs 50K Vitamin D2; Test type: Superiority or Other; p = 0.6, ANOVA

3. Secondary Outcome: Insulin Sensitivity by Matsuda Composite
Description: Insulin Sensitivity by Matsuda Composite - index of insulin sensitivity, higher index means higher insulin sensitivity. Low insulin sensitivity means high insulin resistance and high risk of type 2 diabetes mellitus. It is calculated by a special formula using insulin and glucose measured in Oral Glucose Tolerance test. The formula is different from a formula for OGIS.
  Matsuda composite calculated based on formula 10^4/Square Root of [(fasting glucose x fasting insulin) x (mean glucose x mean insulin)] (Matsuda M, DeFronzo RA. Insulin sensitivity indices obtained from oral glucose tolerance testing: comparison with the euglycemic glucose clamp. Diabetes Care. 1999;22:1462-1470) Unit of measure is 10000/√[(µU/mL)/(mg/dL)]x[(µU/mL)/(mg/dL)].
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: 10^4/√[(µU/mL)/(mg/dL)x(µU/mL)/(mg/dL)]
Arm/Group | Placebo | 50K Vitamin D2
Number analyzed (Participants) | 86 | 87
10^4/√[(µU/mL)/(mg/dL)x(µU/mL)/(mg/dL)] | 0.13 (1.43) | 0.44 (1.51)
Statistical Analysis 1: Comparison: Placebo vs 50K Vitamin D2; Test type: Superiority or Other; p = 0.389, ANOVA

4. Secondary Outcome: Insulinogenic Index-30
Description: Index of insulin secretion, higher index means higher insulin secretion. It is calculated by a special formula using insulin and glucose measured at 0 min and at 30 min (hence 30 in the name) in Oral Glucose Tolerance test.
  Insulin secretion was assessed based on formula Insulinogenic index-30 [(insulin at 30 min - fasting insulin)/(glucose at 30 min - fasting glucose)] (Kosaka K, Hagura R, Kuzuya T. Insulin responses in equivocal and definite diabetes, with special reference to subjects who had mild glucose intolerance but later developed definite diabetes. Diabetes. 1977;26:944-952)
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: (µU/mL)/(mg/dL)
Arm/Group | Placebo | 50K Vitamin D2
Number analyzed (Participants) | 86 | 87
(µU/mL)/(mg/dL) | -0.03 (1.10) | 0.26 (1.03)
Statistical Analysis 1: Comparison: Placebo vs 50K Vitamin D2; Test type: Superiority or Other; p = 0.34, ANOVA — P Value for Insulinogenic Index-30 = 0.34

5. Secondary Outcome: C-Peptidogenic Index-30
Description: Index of insulin secretion, higher index means higher insulin secretion. C-peptide circulates in blood in amounts equal to insulin because insulin and C-peptide are linked when first made by the pancreas. C-peptide is more stable in blood than insulin; therefore it can be reliably used to evaluate insulin secretion. It is calculated by a special formula using C-peptide and glucose measured at 0 min and at 30 min (hence 30 in the name) in Oral Glucose Tolerance test.
  Insulin secretion was assessed based on formula C-Peptidogenic index-30 [(C-Peptide at 30 min - fasting C-peptide)/(glucose at 30 min - fasting glucose)]Bergstrom RW, Wahl PW, Leonetti DL, Fujimoto WY. Association of fasting glucose levels with a delayed secretion of insulin after oral glucose in subjects with glucose intolerance. J Clin Endocrinol Metab. 1990;71:1447-1453.)
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: (ng/mL)/(mg/dL)
Arm/Group | Placebo | 50K Vitamin D2
Number analyzed (Participants) | 86 | 87
(ng/mL)/(mg/dL) | -0.64 (15.84) | 5.32 (17.47)
Statistical Analysis 1: Comparison: Placebo vs 50K Vitamin D2; Test type: Superiority or Other; p = 0.22, ANOVA

6. Post Hoc Outcome: Change in Glycemia
Time Frame: 12 Months
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 50K Vitamin D2
Number analyzed (Participants) | 86 | 87
percentage of participants | 8.3 | 31.6
Statistical Analysis 1: Comparison: Placebo vs 50K Vitamin D2; Test type: Superiority or Other; p = 0.13, Chi-squared

7. Secondary Outcome: Incident Diabetes
Time Frame: 12 Months
Measure: Number; unit: participants
Arm/Group | Placebo | 50K Vitamin D2
Number analyzed (Participants) | 86 | 87
participants | 9 | 9
Statistical Analysis 1: Comparison: Placebo vs 50K Vitamin D2; Test type: Superiority or Other; p = 0.869, Chi-squared

ADVERSE EVENTS:
Time Frame: 12 Months
Groups:
- 50K Vitamin D2: Supplement of vitamin D 400 units provided to all subjects in addition get to D2 50K.
Arm/Group | Placebo | 50K Vitamin D2
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/87
Other Adverse Events (participants affected / at risk) | 0/86 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes